CLINICAL TRIAL: NCT03095495
Title: Heated Humidified High Flow Nasal Cannula (HHHFNC) For Acute Moderate to Severe RSV-Bronchiolitis in Infants Younger Than 3 Months Old: Early Versus Rescue
Brief Title: High Flow Nasal Cannula Therapy in Bronchiolitis : Early vs Rescue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hamad Medical Corporation (Industry)
Collaborators: Sidra Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 16036/16
Record Dates: First submitted 2017-03-06; First posted 2017-03-29 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-05

CONDITIONS: Bronchiolitis; Respiratory Syncytial Virus (RSV)
Keywords: Heated Humidified High Flow Nasal Cannula (HHHFNC); Low Flow Nasal Cannula; Bronchiolitis; Respiratory Syncytial Virus (RSV); Respiratory Failure; High Flow Nasal Cannula (HFNC); Lung Diseases, Obstructive
MeSH Terms: conditions — Bronchiolitis; Respiratory Insufficiency; Lung Diseases, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early use of HHHFNC (Experimental): Heated Humidified High Flow Nasal Cannula
  Interventions: Device: Heated Humidified High Flow Nasal Cannula
- Standard Therapy and Rescue HHHFNC (Active Comparator): Low Flow Nasal Cannula only if the patient needs oxygenation and Rescue HHHFNC if the patient needs PICU
  Interventions: Device: Heated Humidified High Flow Nasal Cannula; Device: Standard Therapy (Low Flow Nasal Cannula)

INTERVENTIONS:
Device: Heated Humidified High Flow Nasal Cannula — HHHFNC therapy is a simple to use system that delivers warm and moist air/oxygen mixture at high flow rates that generate positive airway pressure
Device: Standard Therapy (Low Flow Nasal Cannula) — will be used only if the patient needs oxygenation and Rescue HHHFNC will be used if the patient needs PICU
  Arms: Standard Therapy and Rescue HHHFNC

SUMMARY:
The enrolled RSV-bronchiolitis patients will be randomized into two arms , the early HHHFNC group and the standard therapy group with rescue HHHFNC to study the efficacy of this treatment.

DETAILED DESCRIPTION:
Setting:

The study will be conducted between June 2017 and June 2020 in the short stay unit of the Pediatric Emergency Center (PEC) of Hamad General Hospital, the only pediatric emergency facility in the State of Qatar. Infants aged ≤3 months presenting to the unit for treatment of viral bronchiolitis with positive RSV test will be eligible for the study.

Procedure:

Eligible patients will be enrolled after obtaining written consent. For patients who consent, plain chest radiography, and nasopharyngeal swabs will be taken for RSV detection. If the patient has a positive RSV rapid antigen test, patients will be randomized in one of the study arms. Adverse effects in each group will be carefully monitored and documented.

Study Intervention:

Patients will be randomized into two treatment arms

Group 1: Early HHHFNC Group Patients in this group will be treated by using heated humidified high flow oxygen /air via nasal cannula; investigators will keep the patient on HHHFNC until he/she becomes clinically ready for discharge.

Group 2: Standard Therapy and Rescue HHHFNC Group:

patients in this group will be treated by usual therapy,investigators will use low flow nasal cannula oxygen therapy only if oxygenation needed to maintain Oxygen saturation (SpO2) ≥ 92% , if the patient deteriorate and require ICU, rescue HHHFNC will be started before admission to the ICU.

ELIGIBILITY:
Inclusion Criteria:

* Previously healthy infants with age 0-3 months and gestational age ≥30 weeks admitted to the short stay unit with RSV positive bronchiolitis and clinical severity score ≥4 on Wang clinical severity scale.

Exclusion Criteria:

1. Gestational age less than 30 weeks.
2. Previous history of wheezing.
3. Use of steroid within 48 hours of presentation.
4. History of chronic lung disease.
5. Infants admitted directly to ICU.
6. Prior invasive or non-invasive ventilatory support.
7. Tracheostomy.
8. Nasogastric tubes in situ on admission.
9. Upper airway abnormality (like choanal atresia and midfacial anomalies).
10. Immunodeficient children.
11. History of cardiac disease, renal disease or liver disease.
12. History of neuromuscular disorder.

Max Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2018-08-14 (Actual); Primary Completion 2024-05-28 (Actual); Study Completion 2024-05-28 (Actual)

PRIMARY OUTCOMES:
The rate of Pediatric Intensive Care Unit (PICU) admissions | Through study completion, an average of 3 year
  The rate of Pediatric Intensive Care Unit admissions

SECONDARY OUTCOMES:
Mean length of stay (LOS) | Through study completion, an average of 3 year
  Geometric mean length of stay in the short stay unit
Bronchiolitis Severity Score (BSS) | Up to 72 hours
  Bronchiolitis Severity Score at 4, 8, 12, 24, 36, 48, 72 hours
Percentage of revisit, infirmary short-stay and admission to the hospital or PICU | 2 weeks after discharge
  Percentage of revisit, infirmary short-stay and admission to the hospital or PICU for the same illness on follow up for two weeks post discharge
Transcutaneous Partial Pressure of Carbon Dioxide (PtcCO2) | Up to 72 hours
  Transcutaneous Partial Pressure of Carbon Dioxide (PtcCO2) at 4,8,12,24,36,48,72 hours
Percentage of patients who are on the standard therapy arm and required ICU admission, but improved after the rescue HHHFNC in the ED | 1 hour after starting of rescue HHHFNC
  Percentage of patients who are on the standard therapy arm and required ICU admission, but improved after the rescue HHHFNC in the ED

CONTACTS AND LOCATIONS:
Overall Officials: Khalid Alansari, MD, Principal Investigator — Hamad Medical Corporation
Locations (1):
- Alsadd Pediatric Emergency Center, Doha, Qatar

IPD SHARING:
Plan to Share IPD: No